CLINICAL TRIAL: NCT01611467
Title: A Phase 1 Open-Label Study to Evaluate the Metabolism and Excretion of CC-223 and the Effect of Food on the Pharmacokinetics of CC-223 in Healthy Male Adult Subjects
Acronym: AME/FE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CC-223-CP-002
Record Dates: First submitted 2012-05-25; First posted 2012-06-05 (Estimated); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Safety and Pharmacokinetics in Healthy Volunteer Subjects
Keywords: CC-223; safety; tolerability; pharmacokinetic; AME (Absorption, Metabolism, and Excretion); FE (Food Effect)
MeSH Terms: conditions — Mineralocorticoid Excess Syndrome, Apparent | interventions — CC-223

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 20 mg oral CC-223 with microtracer (Experimental): A single 20-mg oral dose of CC-223 capsule containing a microtracer of [14C]-CC-223 solution
  Interventions: Drug: CC-223
- 20 mg oral CC-223 fasting (Experimental): A single 20-mg oral dose of CC-223 tablet under fasting conditions
  Interventions: Drug: CC-223
- 20 mg oral CC-223 fed (Experimental): A single 20-mg oral dose of CC-223 tablet under fed conditions
  Interventions: Drug: CC-223

INTERVENTIONS:
Drug: CC-223 — 20 mg oral CC-223 capsule containing a microtracer of [14C]-CC-223 solution
  Arms: 20 mg oral CC-223 fasting; 20 mg oral CC-223 fed
Drug: CC-223 — 20-mg oral CC-223 tablet under fasting or fed conditions
  Arms: 20 mg oral CC-223 with microtracer

SUMMARY:
Part 1: To characterize the biotransformation and excretion of CC-223 following a single 20-mg oral dose of CC-223 capsule containing a microtracer of [14C]-CC-223 solution in healthy male subjects; and to evaluate the tolerability of CC-223 after a single 20-mg oral dose of CC-223 capsule containing a microtracer of [14C]-CC-223 solution in healthy male adult subjects Part 2: To evaluate the effect of a high-fat meal on the pharmacokinetics (PK) of CC-223 following a single 20-mg oral dose of CC-223 tablet; To evaluate the effect of a high-fat meal on the PK of M1, the principal pharmacologically-active metabolite, following a single 20-mg oral dose of CC-223 tablet; and to evaluate the tolerability of CC-223 after a single 20-mg oral dose of CC-223 tablet in healthy male adult subjects.

DETAILED DESCRIPTION:
This will be a single-center, 2-part, open-label, randomized (Part 1 only), 2-treatment study in healthy adult males (n = 18). Within no more than 28 days (Day -28) prior to the start of Part 1 or Part 2, subjects will undergo routine screening procedures including physical examination, 12-lead electrocardiograms (ECGs), vital signs, clinical laboratory safety tests (serum chemistry, hematology, and urinalysis), serology screen, fasting glucose levels (including HbA1C) and drug and alcohol screen.

In Part 1, subjects (n = 6) will receive Treatment A (Cohort 1) under fasted conditions. Treatment A: A single 20-mg oral dose of CC-223 capsule containing a microtracer of [14C]- CC-223 solution. For Part 1, subjects will be domiciled at the study center from Day -1 until the morning of Day 8. Upon satisfactory safety review and completion of study-related procedures, subjects will be discharged from the study center on the morning of Day 8.

Part 2 will be a 2-period crossover study; in Period 1, subjects (n = 12) will be randomized to receive an oral 20 mg dose of CC-223 (Treatment B) under fed (n = 6) or fasted (n = 6) conditions. In Period 2, subjects will receive Treatment B under converse conditions based on treatment assignment in Period 1 (Cohort 2 or 3). Fed subjects will be served a standard high fat meal (breakfast), or its equivalent, and must be consumed within 30 minutes of serving. Dosing must occur 30 minutes (±5 minutes) after serving a subject breakfast. All subjects will remain fasted until 4 hours post dose. Subjects will be domiciled at the study center from Day -1 until the morning of Day 5 of each period. Subjects will be discharged from the study center on the morning of Day 5 upon satisfactory safety review and completion of study-related procedures. Periods 1 and 2 will be separated by a washout period of at least 7 days (no more than 10 days) from prior dose to the next dose. In certain instances, a longer washout may be acceptable if previously agreed to by the principal investigator (PI) and Celgene.

All subjects will return to the clinic within 7 to 10 days after the day of discharge in Part 1 or Period 2 of Part 2 for follow-up safety assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Must understand and voluntarily sign a written informed consent document (ICD) prior to any study-related procedures being performed and be able to adhere to restrictions and examination schedules.
2. Must be able to communicate with the investigator and clinical staff and to understand and comply with the requirements of the study.
3. Must be a male 18 to 55 years of age (inclusive) at the time of signing the ICD, with a body mass index (BMI) (weight [kg]/(height [m2]) between 18 and 33 kg/m2 (inclusive) and weight between 60 and 100 kg (132 to 220 lbs; inclusive)
4. Must be healthy (at Screening and Day -1) as determined by the investigator on the basis of medical history, physical examination, clinical laboratory safety test results, vital signs, and 12 lead electrocardiograms (ECGs).

   * Vital signs (systolic and diastolic blood pressure, pulse rate, and oral body temperature) will be assessed in the supine position after the subject has rested for at least 5 minutes.
   * Subject must be afebrile (febrile is defined as ≥ 38.5ºC or 101.3 Fahrenheit)
   * Systolic blood pressure in the range of 90 to 140 mmHg, diastolic blood pressure in the range of 60 to 90 mmHg, and pulse rate in the range of 45 to 100 bpm
   * Screening fasting plasma glucose value within the normal limits of the institution and HbA1C < 6%
5. Subjects (with or without vasectomy) must agree to use barrier contraception (ie, latex condom or any non-latex condom not made out of natural [animal] membrane [eg., polyurethane]) and one other method (eg., spermicide) when engaging in sexual activity with woman of child-bearing potential during study conduct, and for 90 days after the last dose of study medication.
6. Must agree to refrain from donating blood or plasma (other than for this study) while participating in this study and for at least 28 days after the last dose of study drug.

Exclusion Criteria:

1. Recent history (ie, within 3 years) of any clinically significant neurological, gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, endocrine, hematological, dermatological, psychological, or other major disorders.
2. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he were to participate in the study, or confounds the ability to interpret data from the study.
3. Use of any prescribed systemic or topical medication within 30 days of the first dose.
4. Use of any non-prescribed systemic or topical medication (including herbal medicines) within 7 days of the first dose administration (with the exception of vitamin/mineral supplements).
5. Subject used any metabolic enzyme inhibitors or inducers (ie, CYP3A inducers and inhibitors or St. John's Wort) within 30 days of the first dose administration.
6. Presence of any surgical or medical conditions possibly affecting drug absorption, distribution, metabolism, and excretion, or plans to have elective or medical procedures during the conduct of the trial.
7. Exposure to an investigational drug (new chemical entity) within 90 days prior to the first dose administration.
8. Donation of blood or plasma within 60 days prior to the first dose administration.
9. History of multiple (ie, 2 or more) drug allergies.
10. Any clinical significant allergic disease (excluding non-active hay fever), excluding non-active seasonal allergies and childhood asthma cleared for at least 3 years
11. History of drug abuse within 2 years prior to first dosing, or positive urine drug screening test due to illicit drugs.
12. History of alcohol abuse within 2 years prior to dosing, or positive alcohol screen.
13. Smokes more than 10 cigarettes, or consumes the equivalent in tobacco, per day.
14. Known to have, or tests positive for, active or chronic hepatitis B or hepatitis C, or human immunodeficiency virus (HIV) antibodies
15. Received vaccination (excluding seasonal flu vaccination) within 90 days of the study drug administration.
16. For Part 1 Only: Prior exposure to radioactive investigational drugs within 6 months prior to check in, and prior exposure to work-related, diagnostic or therapeutic radiation within 12 months prior to check in.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2012-06-01 (Actual); Primary Completion 2012-07-01 (Actual); Study Completion 2012-07-01 (Actual)

PRIMARY OUTCOMES:
Total radioactivity | Up to 8 days
  Total [14C]-radioactivity in whole blood, plasma, urine and feces
Cumulative excretion of radioactivity | Up to 8 days
  Cumulative excretion of Total [14C]-radioactivity (as fraction of radioactive dose) in urine and feces
Total radioactivity ratios | Up to 8 days
  Total [14C]-radioactivity whole blood-to-plasma ratios
Metabolite concentration | Up to 8 days
  Concentration of CC-223 and M1 metabolite (O-desmethyl-CC-223) in plasma, urine, and feces samples collected up to 14 times from the day prior to dosing to 8 days after dosing.
Cmax | Up to 10 days
  Cmax: Maximum observed concentration in plasma
Tmax | Up to 10 days
  Tmax: Time to maximum concentration
AUC | Up to 10 days
  AUC: Area under the plasma concentration-time curve
t1/2 | Up to 10 days
  t1/2: Terminal half-life

SECONDARY OUTCOMES:
Adverse Events | Up to 30 days
  Number of participants with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Maria Palmisano, M.D., Study Director — Celgene Corporation
Locations (1):
- Covance Research Unit, Inc, Madison, Wisconsin, United States